CLINICAL TRIAL: NCT01096680
Title: A Phase 2, Randomized, Double-Blind, Single Center, Parallel Group, Placebo and Active Comparator, Controlled Study to Evaluate the Pharmacodynamic Profile of Single Doses of SPD489 in Healthy Adult Male Subjects Undergoing a Nocturnal Period of Acute Sleep Loss
Brief Title: Pharmacodynamic Profile of SPD489 in Healthy Adult Males Undergoing a Nocturnal Period of Acute Sleep Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SPD489-207
Record Dates: First submitted 2010-03-30; First posted 2010-03-31 (Estimated); Results first posted 2011-06-23 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Sleep Deprivation
MeSH Terms: conditions — Sleep Deprivation | interventions — Lisdexamfetamine Dimesylate; Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- SPD489 20 mg (Experimental)
  Interventions: Drug: SPD489 20 mg
- SPD489 50 mg (Experimental)
  Interventions: Drug: SPD489 50 mg
- SPD489 70 mg (Experimental)
  Interventions: Drug: SPD489 70 mg
- Armodafinil (Active Comparator)
  Interventions: Drug: Armodafinil
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPD489 20 mg — Single oral dose of 20 mg
  Other Names: Vyvanse
  Arms: SPD489 20 mg
Drug: SPD489 50 mg — Single oral dose of 50 mg
  Other Names: Vyvanse
  Arms: SPD489 50 mg
Drug: SPD489 70 mg — Single oral dose of 70 mg
  Other Names: Vyvanse
  Arms: SPD489 70 mg
Drug: Armodafinil — Single oral dose of 250 mg
  Arms: Armodafinil
Drug: Placebo — Single oral dose
  Arms: Placebo

SUMMARY:
This is a double-blind, single center, parallel group, placebo and active comparator, controlled study to characterize the wake promoting effects of single doses of SPD489 in healthy adult male undergoing acute sleep deprivation.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects between the ages of 18-40 years.
* The subject is in good health and must have a satisfactory medical assessment with no clinically significant and relevant abnormalities (of medical history, physical examination, electrocardiogram (ECG), clinical laboratory evaluation (hematology, biochemistry, and urinalysis).
* Subject has a history of regular sleep-wake habits, routinely spending 6.5-8 hours in bed nightly, and does not oversleep by more than 3 hours on weekends.
* Subject has the ability to provide written, signed, and dated (personally) informed consent to participate in the study, in accordance with the International Conference on Harmonisation Good Clinical Practice Guideline E6 and applicable regulations, before completing any study-related procedures.

Exclusion Criteria:

* Current or relevant previous history of serious, severe, or unstable (acute or progressive) physical or psychiatric illness, any medical disorder that may require treatment or make this subject unlikely to fully complete the study, or any condition that presents undue risk from SPD489 or armodafinil or procedures. Comorbid psychiatric diagnosis will be established by a psychiatric evaluation that includes the Mini International Neuropsychiatric Interview (MINI)-Plus.
* Subject is currently considered a suicide risk, has previously made a suicide attempt, or has a prior history of, or is currently demonstrating suicidal ideation.
* Subject has a known or suspected sleep disorder, or another disorder associated with excessive daytime sleepiness, or any other diagnosis that would interfere with assessing sleepiness in subjects with study related induced sleepiness or abnormal findings on the initial PSG conducted on Day -1 such as, but not limited to, Apnea-Hypopnea Index (AHI) or Periodic Limb Movement Arousal Index (PLMAI) >10.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 135 (Actual)
Dates: Start 2010-04-05 (Actual); Primary Completion 2010-07-18 (Actual); Study Completion 2010-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Clinilabs, Inc., New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- SPD489 20 mg: A single 20 mg oral dose administered (at approximately 7:25pm) prior to a nocturnal period of sleep deprivation
- SPD489 50 mg: A single 50 mg oral dose administered (at approximately 7:25pm) prior to a nocturnal period of sleep deprivation
- SPD489 70 mg: A single 70 mg oral dose administered (at approximately 7:25pm) prior to a nocturnal period of sleep deprivation
- Armodafinil 250 mg: A single 250 mg oral dose administered (at approximately 7:25pm) prior to a nocturnal period of sleep deprivation
- Placebo: A single oral dose of placebo administered (at approximately 7:25pm) prior to a nocturnal period of sleep deprivation
Period: Overall Study
Arm/Group | SPD489 20 mg | SPD489 50 mg | SPD489 70 mg | Armodafinil 250 mg | Placebo
Started | 27 | 27 | 27 | 27 | 27
Completed | 27 | 27 | 27 | 27 | 27
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SPD489 20 mg | SPD489 50 mg | SPD489 70 mg | Armodafinil 250 mg | Placebo | Total
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.4 (5.03) | 28.7 (5.95) | 28.3 (5.04) | 27.0 (5.09) | 28.1 (6.83) | 27.7 (5.62)
Age, Customized [Count of Participants; unit: Participants]
  18 to 40 years | 27 | 27 | 27 | 27 | 27 | 135
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 27 | 27 | 27 | 27 | 27 | 135
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27 | 27 | 27 | 27 | 27 | 135

OUTCOME MEASURES:

1. Primary Outcome: Maintenance of Wakefulness Test (MWT)
Description: The MWT was conducted to determine the subjects' ability to stay awake. Subjects sat in a darkened room and were told to "stay awake as long as possible" during the 30 minute session. This is an indicator of how well you are able to function and remain alert in quiet times of inactivity. Higher times are better.
Time Frame: Over a period of 8 hours
Population: Full Analysis Set (FAS) is defined as all randomized subjects with any primary efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | SPD489 20 mg | SPD489 50 mg | SPD489 70 mg | Armodafinil 250 mg | Placebo
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27
Minutes | 23.3 (1.10) | 27.9 (0.64) | 29.3 (0.44) | 27.6 (0.63) | 15.3 (1.00)
Statistical Analysis 1: Comparison: SPD489 20 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 8.0, 95% CI 2-sided [5.0 to 10.9]
Statistical Analysis 2: Comparison: SPD489 50 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 12.6, 95% CI 2-sided [10.2 to 15.0]
Statistical Analysis 3: Comparison: SPD489 70 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 14.0, 95% CI 2-sided [11.7 to 16.2]
Statistical Analysis 4: Comparison: Armodafinil 250 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 12.3, 95% CI 2-sided [9.9 to 14.7]
Statistical Analysis 5: Comparison: SPD489 20 mg vs Armodafinil 250 mg; Test type: Superiority or Other; p = 0.0014, Mixed Models Analysis; Mean Difference (Final Values) = -4.3, 95% CI 2-sided [-6.9 to -1.8]
Statistical Analysis 6: Comparison: SPD489 50 mg vs Armodafinil 250 mg; Test type: Superiority or Other; p = 0.7601, Mixed Models Analysis; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-1.5 to 2.1]
Statistical Analysis 7: Comparison: SPD489 70 mg vs Armodafinil 250 mg; Test type: Superiority or Other; p = 0.0351, Mixed Models Analysis; Mean Difference (Final Values) = 1.7, 95% CI 2-sided [0.1 to 3.2]

2. Secondary Outcome: Karolinska Sleepiness Scale (KSS) Scores
Description: The KSS is a 9-point scale on which the subject rates sleepiness from 1 (very alert) to 9 (very sleepy/fighting sleep). Lower score is better.
Time Frame: Over a period of 15 hours
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | SPD489 20 mg | SPD489 50 mg | SPD489 70 mg | Armodafinil 250 mg | Placebo
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27
Units on a scale | 4.7 (0.21) | 4.0 (0.21) | 3.6 (0.21) | 4.7 (0.21) | 5.2 (0.21)
Statistical Analysis 1: Comparison: SPD489 20 mg vs Placebo; Test type: Superiority or Other; p = 0.1123, Mixed Models Analysis; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.1 to 0.1]
Statistical Analysis 2: Comparison: SPD489 50 mg vs Placebo; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-1.8 to -0.6]
Statistical Analysis 3: Comparison: SPD489 70 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-2.2 to -1.0]
Statistical Analysis 4: Comparison: Armodafinil 250 mg vs Placebo; Test type: Superiority or Other; p = 0.0947, Mixed Models Analysis; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.1 to 0.1]
Statistical Analysis 5: Comparison: SPD489 20 mg vs Armodafinil 250 mg; Test type: Superiority or Other; p = 0.9393, Mixed Models Analysis; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.6 to 0.6]
Statistical Analysis 6: Comparison: SPD489 50 mg vs Armodafinil 250 mg; Test type: Superiority or Other; p = 0.0297, Mixed Models Analysis; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.3 to -0.1]
Statistical Analysis 7: Comparison: SPD489 70 mg vs Armodafinil 250 mg; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-1.7 to -0.5]

3. Secondary Outcome: KSS Scores by Timepoint
Description: as for outcome 2
Time Frame: Over a period of 15 hours
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | SPD489 20 mg | SPD489 50 mg | SPD489 70 mg | Armodafinil 250 mg | Placebo
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27
Units on a scale
  7:50pm | 2.9 (0.19) | 3.0 (0.19) | 2.6 (0.19) | 2.6 (0.19) | 2.8 (0.19)
  8:50pm | 2.7 (0.20) | 2.7 (0.20) | 2.6 (0.20) | 2.7 (0.20) | 3.0 (0.20)
  9:50pm | 2.9 (0.23) | 3.1 (0.23) | 2.6 (0.23) | 3.1 (0.23) | 3.1 (0.23)
  10:50pm | 2.8 (0.26) | 3.2 (0.26) | 2.4 (0.27) | 2.9 (0.26) | 3.7 (0.27)
  11:50pm | 3.2 (0.29) | 3.1 (0.29) | 2.5 (0.29) | 3.4 (0.29) | 3.9 (0.29)
  12:50am | 3.6 (0.29) | 2.9 (0.29) | 2.6 (0.29) | 3.3 (0.29) | 4.5 (0.29)
  1:50am | 4.0 (0.31) | 3.2 (0.31) | 3.0 (0.31) | 3.8 (0.31) | 4.7 (0.31)
  2:50am | 4.5 (0.35) | 3.7 (0.35) | 3.5 (0.35) | 4.7 (0.35) | 5.7 (0.35)
  3:50am | 5.2 (0.36) | 3.9 (0.36) | 3.7 (0.36) | 5.5 (0.36) | 6.4 (0.36)
  4:50am | 6.1 (0.36) | 4.4 (0.36) | 4.2 (0.36) | 6.0 (0.36) | 6.6 (0.36)
  5:50am | 6.7 (0.37) | 5.1 (0.37) | 4.6 (0.37) | 6.3 (0.37) | 7.1 (0.37)
  6:50am | 6.7 (0.38) | 5.7 (0.38) | 4.8 (0.38) | 6.7 (0.38) | 7.3 (0.38)
  7:50am | 6.5 (0.39) | 5.5 (0.39) | 4.7 (0.39) | 6.6 (0.39) | 7.2 (0.39)
  8:50am | 5.9 (0.41) | 5.0 (0.41) | 4.4 (0.41) | 6.0 (0.41) | 5.4 (0.41)
  9:50am | 5.6 (0.38) | 4.6 (0.38) | 4.5 (0.38) | 5.7 (0.38) | 5.9 (0.38)
  10:50am | 6.2 (0.41) | 5.4 (0.41) | 5.0 (0.41) | 6.0 (0.41) | 6.2 (0.41)
Statistical Analysis 1: Comparison: SPD489 20 mg vs Placebo; 7:50pm; Test type: Superiority or Other; p = 0.7758, Mixed Models Analysis; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.5 to 0.6]
Statistical Analysis 2: Comparison: SPD489 20 mg vs Armodafinil 250 mg; 7:50pm; Test type: Superiority or Other; p = 0.1798, Mixed Models Analysis; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.2 to 0.9]
Statistical Analysis 3: Comparison: SPD489 50 mg vs Placebo; 7:50pm; Test type: Superiority or Other; p = 0.6090, Mixed Models Analysis; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.4 to 0.7]
Statistical Analysis 4: Comparison: SPD489 50 mg vs Armodafinil 250 mg; 7:50pm; Test type: Superiority or Other; p = 0.1169, Mixed Models Analysis; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.1 to 1.0]
Statistical Analysis 5: Comparison: SPD489 70 mg vs Placebo; 7:50pm; Test type: Superiority or Other; p = 0.3028, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.8 to 0.3]
Statistical Analysis 6: Comparison: SPD489 70 mg vs Armodafinil 250 mg; 7:50pm; Test type: Superiority or Other; p = 0.9831, Mixed Models Analysis; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.5 to 0.5]
Statistical Analysis 7: Comparison: Armodafinil 250 mg vs Placebo; 7:50pm; Test type: Superiority or Other; p = 0.2887, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.8 to 0.2]
Statistical Analysis 8: Comparison: SPD489 20 mg vs Placebo; 8:50pm; Test type: Superiority or Other; p = 0.4395, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.8 to 0.3]
Statistical Analysis 9: Comparison: SPD489 20 mg vs Armodafinil 250 mg; 8:50pm; Test type: Superiority or Other; p = 0.9019, Mixed Models Analysis; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.5 to 0.6]
Statistical Analysis 10: Comparison: SPD489 50 mg vs Placebo; 8:50pm; Test type: Superiority or Other; p = 0.3419, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.8 to 0.3]
Statistical Analysis 11: Comparison: SPD489 50 mg vs Armodafinil 250 mg; 8:50pm; Test type: Superiority or Other; p = 0.9581, Mixed Models Analysis; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.6 to 0.5]
Statistical Analysis 12: Comparison: SPD489 70 mg vs Placebo; 8:50pm; Test type: Superiority or Other; p = 0.2572, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.9 to 0.2]
Statistical Analysis 13: Comparison: SPD489 70 mg vs Armodafinil 250 mg; 8:50pm; Test type: Superiority or Other; p = 0.8085, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.6 to 0.5]
Statistical Analysis 14: Comparison: Armodafinil 250 mg vs Placebo; 8:50pm; Test type: Superiority or Other; p = 0.3678, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.8 to 0.3]
Statistical Analysis 15: Comparison: SPD489 20 mg vs Placebo; 9:50pm; Test type: Superiority or Other; p = 0.3732, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.9 to 0.4]
Statistical Analysis 16: Comparison: SPD489 20 mg vs Armodafinil 250 mg; 9:50pm; Test type: Superiority or Other; p = 0.4924, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.9 to 0.4]
Statistical Analysis 17: Comparison: SPD489 50 mg vs Placebo; 9:50pm; Test type: Superiority or Other; p = 0.9798, Mixed Models Analysis; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.7 to 0.6]
Statistical Analysis 18: Comparison: SPD489 50 mg vs Armodafinil 250 mg; 9:50pm; Test type: Superiority or Other; p = 0.8557, Mixed Models Analysis; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.6 to 0.7]
Statistical Analysis 19: Comparison: SPD489 70 mg vs Placebo; 9:50pm; Test type: Superiority or Other; p = 0.0998, Mixed Models Analysis; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.2 to 0.1]
Statistical Analysis 20: Comparison: SPD489 70 mg vs Armodafinil 250 mg; 9:50pm; Test type: Superiority or Other; p = 0.1479, Mixed Models Analysis; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.1 to 0.2]
Statistical Analysis 21: Comparison: Armodafinil 250 mg vs Placebo; 9:50pm; Test type: Superiority or Other; p = 0.8358, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.7 to 0.6]
Statistical Analysis 22: Comparison: SPD489 20 mg vs Placebo; 10:50pm; Test type: Superiority or Other; p = 0.0199, Mixed Models Analysis; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.6 to -0.1]
Statistical Analysis 23: Comparison: SPD489 20 mg vs Armodafinil 250 mg; 10:50pm; Test type: Superiority or Other; p = 0.7625, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.9 to 0.6]
Statistical Analysis 24: Comparison: SPD489 50 mg vs Placebo; 10:50pm; Test type: Superiority or Other; p = 0.1936, Mixed Models Analysis; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.2 to 0.3]
Statistical Analysis 25: Comparison: SPD489 50 mg vs Armodafinil 250 mg; 10:50pm; Test type: Superiority or Other; p = 0.4534, Mixed Models Analysis; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.5 to 1.0]
Statistical Analysis 26: Comparison: SPD489 70 mg vs Placebo; 10:50pm; Test type: Superiority or Other; p = 0.0012, Mixed Models Analysis; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.0 to -0.5]
Statistical Analysis 27: Comparison: SPD489 70 mg vs Armodafinil 250 mg; 10:50pm; Test type: Superiority or Other; p = 0.2072, Mixed Models Analysis; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.2 to 0.3]
Statistical Analysis 28: Comparison: Armodafinil 250 mg vs Placebo; 10:50pm; Test type: Superiority or Other; p = 0.0413, Mixed Models Analysis; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.5 to 0.0]
Statistical Analysis 29: Comparison: SPD489 20 mg vs Placebo; 11:50pm; Test type: Superiority or Other; p = 0.1086, Mixed Models Analysis; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.5 to 0.1]
Statistical Analysis 30: Comparison: SPD489 20 mg vs Armodafinil 250 mg; 11:50pm; Test type: Superiority or Other; p = 0.5843, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-1.0 to 0.6]
Statistical Analysis 31: Comparison: SPD489 50 mg vs Placebo; 11:50pm; Test type: Superiority or Other; p = 0.0571, Mixed Models Analysis; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.6 to 0.0]
Statistical Analysis 32: Comparison: SPD489 50 mg vs Armodafinil 250 mg; 11:50pm; Test type: Superiority or Other; p = 0.3965, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.2 to 0.5]
Statistical Analysis 33: Comparison: SPD489 70 mg vs Placebo; 11:50pm; Test type: Superiority or Other; p = 0.0009, Mixed Models Analysis; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-2.2 to -0.6]
Statistical Analysis 34: Comparison: SPD489 70 mg vs Armodafinil 250 mg; 11:50pm; Test type: Superiority or Other; p = 0.0211, Mixed Models Analysis; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-1.8 to -0.1]
Statistical Analysis 35: Comparison: Armodafinil 250 mg vs Placebo; 11:50pm; Test type: Superiority or Other; p = 0.2863, Mixed Models Analysis; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.2 to 0.4]
Statistical Analysis 36: Comparison: SPD489 20 mg vs Placebo; 12:50am; Test type: Superiority or Other; p = 0.0428, Mixed Models Analysis; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.7 to 0.0]
Statistical Analysis 37: Comparison: SPD489 20 mg vs Armodafinil 250 mg; 12:50am; Test type: Superiority or Other; p = 0.3757, Mixed Models Analysis; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.5 to 1.2]
Statistical Analysis 38: Comparison: SPD489 50 mg vs Placebo; 12:50am; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-2.4 to -0.8]
Statistical Analysis 39: Comparison: SPD489 50 mg vs Armodafinil 250 mg; 12:50am; Test type: Superiority or Other; p = 0.3535, Mixed Models Analysis; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.2 to 0.4]
Statistical Analysis 40: Comparison: SPD489 70 mg vs Placebo; 12:50am; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-2.7 to -1.1]
Statistical Analysis 41: Comparison: SPD489 70 mg vs Armodafinil 250 mg; 12:50am; Test type: Superiority or Other; p = 0.1131, Mixed Models Analysis; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.5 to 0.2]
Statistical Analysis 42: Comparison: Armodafinil 250 mg vs Placebo; 12:50am; Test type: Superiority or Other; p = 0.0039, Mixed Models Analysis; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.0 to -0.4]
Statistical Analysis 43: Comparison: SPD489 20 mg vs Placebo; 1:50am; Test type: Superiority or Other; p = 0.1302, Mixed Models Analysis; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.5 to 0.2]
Statistical Analysis 44: Comparison: SPD489 20 mg vs Armodafinil 250 mg; 1:50am; Test type: Superiority or Other; p = 0.6138, Mixed Models Analysis; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.6 to 1.1]
Statistical Analysis 45: Comparison: SPD489 50 mg vs Placebo; 1:50am; Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-2.3 to -0.6]
Statistical Analysis 46: Comparison: SPD489 50 mg vs Armodafinil 250 mg; 1:50am; Test type: Superiority or Other; p = 0.1643, Mixed Models Analysis; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.5 to 0.3]
Statistical Analysis 47: Comparison: SPD489 70 mg vs Placebo; 1:50am; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-2.5 to -0.8]
Statistical Analysis 48: Comparison: SPD489 70 mg vs Armodafinil 250 mg; 1:50am; Test type: Superiority or Other; p = 0.0782, Mixed Models Analysis; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.6 to 0.1]
Statistical Analysis 49: Comparison: Armodafinil 250 mg vs Placebo; 1:50am; Test type: Superiority or Other; p = 0.0441, Mixed Models Analysis; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.7 to 0.0]
Statistical Analysis 50: Comparison: SPD489 20 mg vs Placebo; 2:50am; Test type: Superiority or Other; p = 0.0193, Mixed Models Analysis; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.2 to -0.2]
Statistical Analysis 51: Comparison: SPD489 20 mg vs Armodafinil 250 mg; 2:50am; Test type: Superiority or Other; p = 0.7071, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-1.2 to 0.8]
Statistical Analysis 52: Comparison: SPD489 50 mg vs Placebo; 2:50am; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-2.9 to -0.9]
Statistical Analysis 53: Comparison: SPD489 50 mg vs Armodafinil 250 mg; 2:50am; Test type: Superiority or Other; p = 0.0611, Mixed Models Analysis; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.9 to 0.0]
Statistical Analysis 54: Comparison: SPD489 70 mg vs Placebo; 2:50am; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-3.2 to -1.2]
Statistical Analysis 55: Comparison: SPD489 70 mg vs Armodafinil 250 mg; 2:50am; Test type: Superiority or Other; p = 0.0160, Mixed Models Analysis; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.2 to -0.2]
Statistical Analysis 56: Comparison: Armodafinil 250 mg vs Placebo; 2:50am; Test type: Superiority or Other; p = 0.0480, Mixed Models Analysis; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-2.0 to 0.0]
Statistical Analysis 57: Comparison: SPD489 20 mg vs Placebo; 3:50am; Test type: Superiority or Other; p = 0.0234, Mixed Models Analysis; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.2 to -0.2]
Statistical Analysis 58: Comparison: SPD489 20 mg vs Armodafinil 250 mg; 3:50am; Test type: Superiority or Other; p = 0.5624, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.3 to 0.7]
Statistical Analysis 59: Comparison: SPD489 50 mg vs Placebo; 3:50am; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-3.5 to -1.5]
Statistical Analysis 60: Comparison: SPD489 50 mg vs Armodafinil 250 mg; 3:50am; Test type: Superiority or Other; p = 0.0022, Mixed Models Analysis; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-2.6 to -0.6]
Statistical Analysis 61: Comparison: SPD489 70 mg vs Placebo; 3:50am; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -2.7, 95% CI 2-sided [-3.7 to -1.6]
Statistical Analysis 62: Comparison: SPD489 70 mg vs Armodafinil 250 mg; 3:50am; Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-2.8 to -0.8]
Statistical Analysis 63: Comparison: Armodafinil 250 mg vs Placebo; 3:50am; Test type: Superiority or Other; p = 0.0883, Mixed Models Analysis; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.9 to 0.1]
Statistical Analysis 64: Comparison: SPD489 20 mg vs Placebo; 4:50am; Test type: Superiority or Other; p = 0.3093, Mixed Models Analysis; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.5 to 0.5]
Statistical Analysis 65: Comparison: SPD489 20 mg vs Armodafinil 250 mg; 4:50am; Test type: Superiority or Other; p = 0.8871, Mixed Models Analysis; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.9 to 1.1]
Statistical Analysis 66: Comparison: SPD489 50 mg vs Placebo; 4:50am; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-3.2 to -1.2]
Statistical Analysis 67: Comparison: SPD489 50 mg vs Armodafinil 250 mg; 4:50am; Test type: Superiority or Other; p = 0.0022, Mixed Models Analysis; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-2.6 to -0.6]
Statistical Analysis 68: Comparison: SPD489 70 mg vs Placebo; 4:50am; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-3.4 to -1.4]
Statistical Analysis 69: Comparison: SPD489 70 mg vs Armodafinil 250 mg; 4:50am; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-2.8 to -0.8]
Statistical Analysis 70: Comparison: Armodafinil 250 mg vs Placebo; 4:50am; Test type: Superiority or Other; p = 0.2462, Mixed Models Analysis; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.6 to 0.4]
Statistical Analysis 71: Comparison: SPD489 20 mg vs Placebo; 5:50am; Test type: Superiority or Other; p = 0.4427, Mixed Models Analysis; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.4 to 0.6]
Statistical Analysis 72: Comparison: SPD489 20 mg vs Armodafinil 250 mg; 5:50am; Test type: Superiority or Other; p = 0.4405, Mixed Models Analysis; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.6 to 1.4]
Statistical Analysis 73: Comparison: SPD489 50 mg vs Placebo; 5:50am; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-3.0 to -0.9]
Statistical Analysis 74: Comparison: SPD489 50 mg vs Armodafinil 250 mg; 5:50am; Test type: Superiority or Other; p = 0.0279, Mixed Models Analysis; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.2 to -0.1]
Statistical Analysis 75: Comparison: SPD489 70 mg vs Placebo; 5:50am; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-3.5 to -1.5]
Statistical Analysis 76: Comparison: SPD489 70 mg vs Armodafinil 250 mg; 5:50am; Test type: Superiority or Other; p = 0.0015, Mixed Models Analysis; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-2.7 to -0.7]
Statistical Analysis 77: Comparison: Armodafinil 250 mg vs Placebo; 5:50am; Test type: Superiority or Other; p = 0.1246, Mixed Models Analysis; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.8 to 0.2]
Statistical Analysis 78: Comparison: SPD489 20 mg vs Placebo; 6:50am; Test type: Superiority or Other; p = 0.3067, Mixed Models Analysis; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.6 to 0.5]
Statistical Analysis 79: Comparison: SPD489 20 mg vs Armodafinil 250 mg; 6:50am; Test type: Superiority or Other; p = 0.8940, Mixed Models Analysis; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-1.0 to 1.1]
Statistical Analysis 80: Comparison: SPD489 50 mg vs Placebo; 6:50am; Test type: Superiority or Other; p = 0.0034, Mixed Models Analysis; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-2.7 to -0.5]
Statistical Analysis 81: Comparison: SPD489 50 mg vs Armodafinil 250 mg; 6:50am; Test type: Superiority or Other; p = 0.0708, Mixed Models Analysis; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-2.0 to 0.1]
Statistical Analysis 82: Comparison: SPD489 70 mg vs Placebo; 6:50am; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-3.6 to -1.4]
Statistical Analysis 83: Comparison: SPD489 70 mg vs Armodafinil 250 mg; 6:50am; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-2.9 to -0.8]
Statistical Analysis 84: Comparison: Armodafinil 250 mg vs Placebo; 6:50am; Test type: Superiority or Other; p = 0.2476, Mixed Models Analysis; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.7 to 0.4]
Statistical Analysis 85: Comparison: SPD489 20 mg vs Placebo; 7:50am; Test type: Superiority or Other; p = 0.2310, Mixed Models Analysis; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.8 to 0.4]
Statistical Analysis 86: Comparison: SPD489 20 mg vs Armodafinil 250 mg; 7:50am; Test type: Superiority or Other; p = 0.8369, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-1.2 to 1.0]
Statistical Analysis 87: Comparison: SPD489 50 mg vs Placebo; 7:50am; Test type: Superiority or Other; p = 0.0035, Mixed Models Analysis; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-2.7 to -0.5]
Statistical Analysis 88: Comparison: SPD489 50 mg vs Armodafinil 250 mg; 7:50am; Test type: Superiority or Other; p = 0.0498, Mixed Models Analysis; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-2.2 to 0.0]
Statistical Analysis 89: Comparison: SPD489 70 mg vs Placebo; 7:50am; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-3.6 to -1.4]
Statistical Analysis 90: Comparison: SPD489 70 mg vs Armodafinil 250 mg; 7:50am; Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-3.0 to -0.8]
Statistical Analysis 91: Comparison: Armodafinil 250 mg vs Placebo; 7:50am; Test type: Superiority or Other; p = 0.3198, Mixed Models Analysis; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.6 to 0.5]
Statistical Analysis 92: Comparison: SPD489 20 mg vs Placebo; 8:50am; Test type: Superiority or Other; p = 0.3750, Mixed Models Analysis; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-0.6 to 1.7]
Statistical Analysis 93: Comparison: SPD489 20 mg vs Armodafinil 250 mg; 8:50am; Test type: Superiority or Other; p = 0.7978, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-1.3 to 1.0]
Statistical Analysis 94: Comparison: SPD489 50 mg vs Placebo; 8:50am; Test type: Superiority or Other; p = 0.5197, Mixed Models Analysis; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.5 to 0.8]
Statistical Analysis 95: Comparison: SPD489 50 mg vs Armodafinil 250 mg; 8:50am; Test type: Superiority or Other; p = 0.0751, Mixed Models Analysis; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-2.2 to 0.1]
Statistical Analysis 96: Comparison: SPD489 70 mg vs Placebo; 8:50am; Test type: Superiority or Other; p = 0.1079, Mixed Models Analysis; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-2.1 to 0.2]
Statistical Analysis 97: Comparison: SPD489 70 mg vs Armodafinil 250 mg; 8:50am; Test type: Superiority or Other; p = 0.0065, Mixed Models Analysis; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-2.8 to -0.5]
Statistical Analysis 98: Comparison: Armodafinil 250 mg vs Placebo; 8:50am; Test type: Superiority or Other; p = 0.2529, Mixed Models Analysis; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-0.5 to 1.8]
Statistical Analysis 99: Comparison: SPD489 20 mg vs Placebo; 9:50am; Test type: Superiority or Other; p = 0.6364, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.3 to 0.8]
Statistical Analysis 100: Comparison: SPD489 20 mg vs Armodafinil 250 mg; 9:50am; Test type: Superiority or Other; p = 0.9417, Mixed Models Analysis; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-1.1 to 1.0]
Statistical Analysis 101: Comparison: SPD489 50 mg vs Placebo; 9:50am; Test type: Superiority or Other; p = 0.0200, Mixed Models Analysis; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-2.3 to -0.2]
Statistical Analysis 102: Comparison: SPD489 50 mg vs Armodafinil 250 mg; 9:50am; Test type: Superiority or Other; p = 0.0527, Mixed Models Analysis; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-2.1 to 0.0]
Statistical Analysis 103: Comparison: SPD489 70 mg vs Placebo; 9:50am; Test type: Superiority or Other; p = 0.0107, Mixed Models Analysis; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-2.5 to -0.3]
Statistical Analysis 104: Comparison: SPD489 70 mg vs Armodafinil 250 mg; 9:50am; Test type: Superiority or Other; p = 0.0303, Mixed Models Analysis; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.2 to -0.1]
Statistical Analysis 105: Comparison: Armodafinil 250 mg vs Placebo; 9:50am; Test type: Superiority or Other; p = 0.6889, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-1.3 to 0.8]
Statistical Analysis 106: Comparison: SPD489 20 mg vs Placebo; 10:50am; Test type: Superiority or Other; p = 0.9552, Mixed Models Analysis; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-1.2 to 1.1]
Statistical Analysis 107: Comparison: SPD489 20 mg vs Armodafinil 250 mg; 10:50am; Test type: Superiority or Other; p = 0.7558, Mixed Models Analysis; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-1.0 to 1.3]
Statistical Analysis 108: Comparison: SPD489 50 mg vs Placebo; 10:50am; Test type: Superiority or Other; p = 0.1824, Mixed Models Analysis; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.9 to 0.4]
Statistical Analysis 109: Comparison: SPD489 50 mg vs Armodafinil 250 mg; 10:50am; Test type: Superiority or Other; p = 0.3323, Mixed Models Analysis; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.7 to 0.6]
Statistical Analysis 110: Comparison: SPD489 70 mg vs Placebo; 10:50am; Test type: Superiority or Other; p = 0.0413, Mixed Models Analysis; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.4 to 0.0]
Statistical Analysis 111: Comparison: SPD489 70 mg vs Armodafinil 250 mg; 10:50am; Test type: Superiority or Other; p = 0.0925, Mixed Models Analysis; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-2.2 to 0.2]
Statistical Analysis 112: Comparison: Armodafinil 250 mg vs Placebo; 10:50am; Test type: Superiority or Other; p = 0.7133, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-1.4 to 0.9]

4. Secondary Outcome: Psychomotor Vigilance Task (PVT) Scores
Description: PVT assesses behavioral alertness. Subjects were required to respond to a visual stimulus by pressing a button on a mechanical device and the reaction time was measured. Higher scores indicate attention lapses.
Time Frame: Over a period of 12 hours
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | SPD489 20 mg | SPD489 50 mg | SPD489 70 mg | Armodafinil 250 mg | Placebo
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27
msec | 243.6 (3.59) | 234.8 (3.58) | 243.5 (3.58) | 243.7 (3.59) | 270.2 (3.59)
Statistical Analysis 1: Comparison: SPD489 20 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -26.5, 95% CI 2-sided [-36.6 to -16.5]
Statistical Analysis 2: Comparison: SPD489 50 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -35.4, 95% CI 2-sided [-45.5 to -25.4]
Statistical Analysis 3: Comparison: SPD489 70 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -26.7, 95% CI 2-sided [-36.7 to -16.6]
Statistical Analysis 4: Comparison: Armodafinil 250 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -26.5, 95% CI 2-sided [-36.6 to -16.5]
Statistical Analysis 5: Comparison: SPD489 20 mg vs Armodafinil 250 mg; Test type: Superiority or Other; p = 0.9945, Mixed Models Analysis; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-10.1 to 10.0]
Statistical Analysis 6: Comparison: SPD489 50 mg vs Armodafinil 250 mg; Test type: Superiority or Other; p = 0.0814, Mixed Models Analysis; Mean Difference (Final Values) = -8.9, 95% CI 2-sided [-18.9 to 1.1]
Statistical Analysis 7: Comparison: SPD489 70 mg vs Armodafinil 250 mg; Test type: Superiority or Other; p = 0.9743, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-10.2 to 9.9]

5. Secondary Outcome: PVT Scores by Timepoint
Description: as for outcome 4
Time Frame: Over a period of 12 hours
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | SPD489 20 mg | SPD489 50 mg | SPD489 70 mg | Armodafinil 250 mg | Placebo
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27
msec
  9:15pm | 231.6 (3.50) | 233.2 (3.49) | 234.9 (3.49) | 235.5 (3.49) | 241.3 (3.50)
  11:15pm | 232.6 (2.98) | 230.9 (2.97) | 231.2 (2.97) | 229.3 (2.97) | 249.3 (2.98)
  1:15am | 231.5 (3.89) | 231.5 (3.88) | 230.2 (3.89) | 233.0 (3.88) | 256.7 (3.89)
  3:15am | 243.6 (4.65) | 227.4 (4.64) | 240.7 (4.64) | 242.5 (4.64) | 280.7 (4.65)
  5:15am | 253.4 (4.67) | 237.7 (4.66) | 242.5 (4.66) | 249.5 (4.66) | 291.6 (4.67)
  7:15am | 257.9 (7.67) | 242.6 (7.67) | 259.2 (7.67) | 259.1 (7.67) | 295.5 (7.67)
  9:15am | 254.8 (10.84) | 240.0 (10.84) | 265.9 (10.84) | 256.7 (10.93) | 276.1 (10.84)
Statistical Analysis 1: Comparison: SPD489 20 mg vs Placebo; 9:15pm; Test type: Superiority or Other; p = 0.0544, Mixed Models Analysis; Mean Difference (Final Values) = -9.6, 95% CI 2-sided [-19.4 to 0.2]
Statistical Analysis 2: Comparison: SPD489 20 mg vs Armodafinil 250 mg; 9:15pm; Test type: Superiority or Other; p = 0.4410, Mixed Models Analysis; Mean Difference (Final Values) = -3.8, 95% CI 2-sided [-13.6 to 6.0]
Statistical Analysis 3: Comparison: SPD489 50 mg vs Placebo; 9:15pm; Test type: Superiority or Other; p = 0.1046, Mixed Models Analysis; Mean Difference (Final Values) = -8.1, 95% CI 2-sided [-17.9 to 1.7]
Statistical Analysis 4: Comparison: SPD489 50 mg vs Armodafinil 250 mg; 9:15pm; Test type: Superiority or Other; p = 0.6467, Mixed Models Analysis; Mean Difference (Final Values) = -2.3, 95% CI 2-sided [-12.0 to 7.5]
Statistical Analysis 5: Comparison: SPD489 70 mg vs Placebo; 9:15pm; Test type: Superiority or Other; p = 0.1971, Mixed Models Analysis; Mean Difference (Final Values) = -6.4, 95% CI 2-sided [-16.2 to 3.4]
Statistical Analysis 6: Comparison: SPD489 70 mg vs Armodafinil 250 mg; 9:15pm; Test type: Superiority or Other; p = 0.9052, Mixed Models Analysis; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-10.4 to 9.2]
Statistical Analysis 7: Comparison: Armodafinil 250 mg vs Placebo; 9:15pm; Test type: Superiority or Other; p = 0.2420, Mixed Models Analysis; Mean Difference (Final Values) = -5.8, 95% CI 2-sided [-15.6 to 4.0]
Statistical Analysis 8: Comparison: SPD489 20 mg vs Placebo; 11:15pm; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -16.7, 95% CI 2-sided [-25.1 to -8.3]
Statistical Analysis 9: Comparison: SPD489 20 mg vs Armodafinil 250 mg; 11:15pm; Test type: Superiority or Other; p = 0.4321, Mixed Models Analysis; Mean Difference (Final Values) = 3.3, 95% CI 2-sided [-5.0 to 11.6]
Statistical Analysis 10: Comparison: SPD489 50 mg vs Placebo; 11:15pm; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -18.4, 95% CI 2-sided [-26.7 to -10.1]
Statistical Analysis 11: Comparison: SPD489 50 mg vs Armodafinil 250 mg; 11:15pm; Test type: Superiority or Other; p = 0.6999, Mixed Models Analysis; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [-6.7 to 9.9]
Statistical Analysis 12: Comparison: SPD489 70 mg vs Placebo; 11:15pm; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -18.1, 95% CI 2-sided [-26.4 to -9.8]
Statistical Analysis 13: Comparison: SPD489 70 mg vs Armodafinil 250 mg; 11:15pm; Test type: Superiority or Other; p = 0.6566, Mixed Models Analysis; Mean Difference (Final Values) = 1.9, 95% CI 2-sided [-6.4 to 10.2]
Statistical Analysis 14: Comparison: Armodafinil 250 mg vs Placebo; 11:15pm; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -20.0, 95% CI 2-sided [-28.3 to -11.7]
Statistical Analysis 15: Comparison: SPD489 20 mg vs Placebo; 1:15am; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -25.2, 95% CI 2-sided [-36.1 to -14.3]
Statistical Analysis 16: Comparison: SPD489 20 mg vs Armodafinil 250 mg; 1:15am; Test type: Superiority or Other; p = 0.7824, Mixed Models Analysis; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-12.4 to 9.4]
Statistical Analysis 17: Comparison: SPD489 50 mg vs Placebo; 1:15am; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -25.1, 95% CI 2-sided [-36.0 to -14.3]
Statistical Analysis 18: Comparison: SPD489 50 mg vs Armodafinil 250 mg; 1:15am; Test type: Superiority or Other; p = 0.7867, Mixed Models Analysis; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-12.4 to 9.4]
Statistical Analysis 19: Comparison: SPD489 70 mg vs Placebo; 1:15am; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -26.5, 95% CI 2-sided [-37.4 to -15.6]
Statistical Analysis 20: Comparison: SPD489 70 mg vs Armodafinil 250 mg; 1:15am; Test type: Superiority or Other; p = 0.6029, Mixed Models Analysis; Mean Difference (Final Values) = -2.9, 95% CI 2-sided [-13.7 to 8.0]
Statistical Analysis 21: Comparison: Armodafinil 250 mg vs Placebo; 1:15am; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -23.6, 95% CI 2-sided [-34.5 to -12.8]
Statistical Analysis 22: Comparison: SPD489 20 mg vs Placebo; 3:15am; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -37.1, 95% CI 2-sided [-50.1 to -24.1]
Statistical Analysis 23: Comparison: SPD489 20 mg vs Armodafinil 250 mg; 3:15am; Test type: Superiority or Other; p = 0.8684, Mixed Models Analysis; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [-11.9 to 14.1]
Statistical Analysis 24: Comparison: SPD489 50 mg vs Placebo; 3:15am; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -53.3, 95% CI 2-sided [-66.3 to -40.3]
Statistical Analysis 25: Comparison: SPD489 50 mg vs Armodafinil 250 mg; 3:15am; Test type: Superiority or Other; p = 0.0228, Mixed Models Analysis; Mean Difference (Final Values) = -15.1, 95% CI 2-sided [-28.1 to -2.1]
Statistical Analysis 26: Comparison: SPD489 70 mg vs Placebo; 3:15am; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -40.0, 95% CI 2-sided [-53.0 to -27.0]
Statistical Analysis 27: Comparison: SPD489 70 mg vs Armodafinil 250 mg; 3:15am; Test type: Superiority or Other; p = 0.7852, Mixed Models Analysis; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-14.8 to 11.2]
Statistical Analysis 28: Comparison: Armodafinil 250 mg vs Placebo; 3:15am; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -38.2, 95% CI 2-sided [-51.2 to -25.2]
Statistical Analysis 29: Comparison: SPD489 20 mg vs Placebo; 5:15am; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -38.2, 95% CI 2-sided [-51.3 to -25.1]
Statistical Analysis 30: Comparison: SPD489 20 mg vs Armodafinil 250 mg; 5:15am; Test type: Superiority or Other; p = 0.5528, Mixed Models Analysis; Mean Difference (Final Values) = 3.9, 95% CI 2-sided [-9.1 to 17.0]
Statistical Analysis 31: Comparison: SPD489 50 mg vs Placebo; 5:15am; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -53.9, 95% CI 2-sided [-67.0 to -40.9]
Statistical Analysis 32: Comparison: SPD489 50 mg vs Armodafinil 250 mg; 5:15am; Test type: Superiority or Other; p = 0.0747, Mixed Models Analysis; Mean Difference (Final Values) = -11.8, 95% CI 2-sided [-24.9 to 1.2]
Statistical Analysis 33: Comparison: SPD489 70 mg vs Placebo; 5:15am; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -49.2, 95% CI 2-sided [-62.2 to -36.1]
Statistical Analysis 34: Comparison: SPD489 70 mg vs Armodafinil 250 mg; 5:15am; Test type: Superiority or Other; p = 0.2868, Mixed Models Analysis; Mean Difference (Final Values) = -7.1, 95% CI 2-sided [-20.1 to 6.0]
Statistical Analysis 35: Comparison: Armodafinil 250 mg vs Placebo; 5:15am; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -42.1, 95% CI 2-sided [-55.2 to -29.1]
Statistical Analysis 36: Comparison: SPD489 20 mg vs Placebo; 7:15am; Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis; Mean Difference (Final Values) = -37.6, 95% CI 2-sided [-59.1 to -16.2]
Statistical Analysis 37: Comparison: SPD489 20 mg vs Armodafinil 250 mg; 7:15am; Test type: Superiority or Other; p = 0.9089, Mixed Models Analysis; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-22.7 to 20.2]
Statistical Analysis 38: Comparison: SPD489 50 mg vs Placebo; 7:15am; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -52.9, 95% CI 2-sided [-74.3 to -31.4]
Statistical Analysis 39: Comparison: SPD489 50 mg vs Armodafinil 250 mg; 7:15am; Test type: Superiority or Other; p = 0.1307, Mixed Models Analysis; Mean Difference (Final Values) = -16.5, 95% CI 2-sided [-37.9 to 5.0]
Statistical Analysis 40: Comparison: SPD489 70 mg vs Placebo; 7:15am; Test type: Superiority or Other; p = 0.0011, Mixed Models Analysis; Mean Difference (Final Values) = -36.3, 95% CI 2-sided [-57.7 to -14.8]
Statistical Analysis 41: Comparison: SPD489 70 mg vs Armodafinil 250 mg; 7:15am; Test type: Superiority or Other; p = 0.9903, Mixed Models Analysis; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-21.3 to 21.6]
Statistical Analysis 42: Comparison: Armodafinil 250 mg vs Placebo; 7:15am; Test type: Superiority or Other; p = 0.0010, Mixed Models Analysis; Mean Difference (Final Values) = -36.4, 95% CI 2-sided [-57.8 to -14.9]
Statistical Analysis 43: Comparison: SPD489 20 mg vs Placebo; 9:15am; Test type: Superiority or Other; p = 0.1655, Mixed Models Analysis; Mean Difference (Final Values) = -21.4, 95% CI 2-sided [-51.7 to 9.0]
Statistical Analysis 44: Comparison: SPD489 20 mg vs Armodafinil 250 mg; 9:15am; Test type: Superiority or Other; p = 0.8975, Mixed Models Analysis; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-32.4 to 28.5]
Statistical Analysis 45: Comparison: SPD489 50 mg vs Placebo; 9:15am; Test type: Superiority or Other; p = 0.0199, Mixed Models Analysis; Mean Difference (Final Values) = -36.2, 95% CI 2-sided [-66.5 to -5.8]
Statistical Analysis 46: Comparison: SPD489 50 mg vs Armodafinil 250 mg; 9:15am; Test type: Superiority or Other; p = 0.2785, Mixed Models Analysis; Mean Difference (Final Values) = -16.8, 95% CI 2-sided [-47.2 to 13.7]
Statistical Analysis 47: Comparison: SPD489 70 mg vs Placebo; 9:15am; Test type: Superiority or Other; p = 0.5048, Mixed Models Analysis; Mean Difference (Final Values) = -10.3, 95% CI 2-sided [-40.6 to 20.1]
Statistical Analysis 48: Comparison: SPD489 70 mg vs Armodafinil 250 mg; 9:15am; Test type: Superiority or Other; p = 0.5533, Mixed Models Analysis; Mean Difference (Final Values) = 9.1, 95% CI 2-sided [-21.3 to 39.6]
Statistical Analysis 49: Comparison: Armodafinil 250 mg vs Placebo; 9:15am; Test type: Superiority or Other; p = 0.2098, Mixed Models Analysis; Mean Difference (Final Values) = -19.4, 95% CI 2-sided [-49.9 to 11.1]

ADVERSE EVENTS:
Description: Safety Analysis Set
Arm/Group | SPD489 20 mg | SPD489 50 mg | SPD489 70 mg | Armodafinil 250 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/27 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 1/27 | 5/27 | 4/27 | 3/27 | 1/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SPD489 20 mg (N=27) | SPD489 50 mg (N=27) | SPD489 70 mg (N=27) | Armodafinil 250 mg (N=27) | Placebo (N=27)
Headache (Nervous system disorders) | 0 | 4 | 2 | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.